CLINICAL TRIAL: NCT01962610
Title: Improving Management of Acute Pain for Older Adults in the ED Setting
Brief Title: Improving Pain Management for Older Adults in the Emergency Department (ED)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: GCO 10-1414; 5R21AG040734-02 (NIH)
Record Dates: First submitted 2013-09-10; First posted 2013-10-14 (Estimated); Last update posted 2015-11-05 (Estimated); Status verified 2015-11

CONDITIONS: Abdominal Pain Care
Keywords: Pain care; emergency; clinical decision support; abdominal pain
MeSH Terms: conditions — Emergencies; Abdominal Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ePCA and Pain keycept intervention (Experimental): Study designed ePCA and pain keycept interventions are embedded in electronic medical record during patient ED visit
  Interventions: Other: ePCA and Pain keycept intervention
- Usual Care (No Intervention): No study designed ePCA and pain keycept interventions are embedded in electronic medical record during patient ED visit

INTERVENTIONS:
Other: ePCA and Pain keycept intervention — Study designed ePCA and pain keycept interventions are embedded in electronic medical record during patient ED visit.
  Arms: ePCA and Pain keycept intervention

SUMMARY:
The goals of this exploratory study are to determine the feasibility of integrating electronic clinical decision support into routine clinical pain care for adults in the ED setting and gather data on whether or not such clinical decision support is effective in improving pain care outcomes in the ED. The use of an electronic pain care alert (ePCA) prompting doctors to provide acute pain care for adult patients with complaints of severe abdominal pain will be compared to patients seen by clinicians with routine ED care.

Hypothesis: The ePCA will improve the quality of acute pain care for patients.

DETAILED DESCRIPTION:
This study will compare the effectiveness of the combined electronic pain care alert (ePCA) and "pain keycepts" (i.e., embedded pain care concepts/algorithms within clinician documentation templates) intervention versus routine care on acute pain care outcomes for geriatric abdominal pain patients in severe pain.

Hypothesis: The ePCA and pain keycept will improve the quality of acute pain care (i.e., Geriatric pain care quality indicators that include improved pain evaluation and pain treatment (better pain assessment documentation, earlier administration of analgesic medication, greater reduction of pain levels)) for geriatric abdominal pain patients in severe pain.

Study Design: This is an exploratory randomized trial of the intervention versus usual clinical care (control).

1. (Pre-intervention abdominal pain care baseline): Prior to any implementation of the ePCA, baseline Epic process of pain care measures for abdominal pain patients will be collected for a 4-month period. Study variables will be collected to determine baseline patient-related and abdominal pain care data. Baseline data will be used for two purposes. To determine if there: 1.) is an improvement in the quality of pain care received post-intervention and 2.) are treatment diffusion effects with the control (routine care) physicians who do not receive ePCAs (i.e., after the intervention period has commenced, are differences in process of pain care outcomes found for the control group versus pre-intervention baseline group).
2. This will be a randomized comparative effectiveness trial gathering pilot data on the efficacy of the ePCA to improve with ED pain care for adults with severe abdominal pain. To study the effect of the ePCA intervention, the alert will be randomized to RESIDENT physicians, who will be randomly assigned to groups designated in the Epic EMR (electronic medical record) (i.e., the alert will be triggered for some residents, and not triggered for other residents (usual care) for the entire study period). Both groups will have equal privileges in all ways (i.e., documentation and ordering) except that BPAs will or will not be integrated for intervention vs. control. Investigators will be blinded to randomization assignments and subjects (resident physicians) will be blinded to study aims. Residents will always remain in their initial randomized arm.

The unit of analysis will be the ED visit. To study the impact of the ePCA on pain care outcomes, pilot data will be collected with prospective survey from abdominal pain patients, automated data reports from Epic and MSDW, and medical record review. Eligible subjects enrolled and consented will be surveyed at discharge from the ED with regard to pain scores, desire for analgesic medication, and satisfaction with pain care. While evidence from the Surgical and Emergency Medicine (EM) literature indicate early analgesia does not obscure clinical diagnoses, not result in diagnostic delays, nor impedes informed consent, some clinicians may withhold analgesia due to the continued misguided belief that analgesia may mask diagnostic findings or invalidate consent. For this reason, data will also be collected of whether or not the patient required surgical consultation.

ELIGIBILITY:
Inclusion Criteria:

Resident physicians will be included if:

* they provide care to adult patients in the Icahn School of Medicine at Mount Sinai's ED.

Patients will be enrolled for survey and/or medical record review if

* All adult (≥20 years) patients seen in the Icahn School of Medicine at Mount Sinai's ED
* with severe pain (≥10 on a verbal pain scale of 0-10, 0=none, 10=severe)
* and chief complaints of abdominal pain will be eligible for retrospective and/or medical record review and prospective survey at ED discharge.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4693 (Actual)
Dates: Start 2011-06; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Analgesia order | at ED visit
  pain care outcomes - analgesic medication ordering status
Analgesia Administration | at ED visit
  pain care outcomes - Times from ED arrival to analgesic medication administration

SECONDARY OUTCOMES:
Patient Pain Care Satisfaction | at ED visit
  Eligible subjects will be surveyed at ED discharge with regard to pain scores, desire for analgesic medication and satisfaction with pain care.

CONTACTS AND LOCATIONS:
Overall Officials: Ula Y Hwang, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Mediciine at Mount Sinai, New York, New York, United States